CLINICAL TRIAL: NCT01492517
Title: Epigenetic Effects of Diesel Exhaust and Ozone Exposure
Acronym: Lamarck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Diaz-Sanchez, Chief, Clinical Research Branch, Environmental Protection Agency (EPA)
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: E10-025CS
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-02

CONDITIONS: Exposure to Pollution; Inhalation of Ozone
Keywords: Controlled Human exposure study; Air Pollution; Gene expression; Epigenetic; Cardiovascular
MeSH Terms: interventions — Vehicle Emissions; 1-(2-(dodecyloxy)ethyl)pyrrolidine hydrochloride; Environment, Controlled

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Clean air exposure (Sham Comparator): Exposure to clean air will be conducted in an exposure chamber at the EPA Human Studies Facility on the UNC campus. Each subject will be exposed to clean air for 2 hours. Subjects will begin exercising on an exercise bike. Each exercise session will consist of a 15 minute exercise interval at a level of up to 25 L/m2/BSA followed by a 15 minute rest period. The exposure atmosphere will be at approximately 40 + 10% RH and approximately 22 + 2 oC.
  Interventions: Other: Clean Air
- Ozone exposure (Other): Exposure to 0.3ppm ozone will be conducted in an exposure chamber at the EPA Human Studies Facility on the UNC campus. Each subject will be exposed for 2 hours. Subjects will begin exercising on an exercise bike. Each exercise session will consist of a 15 minute exercise interval at a level of up to 25 L/m2/BSA followed by a 15 minute rest period. The exposure atmosphere will be at approximately 40 + 10% RH and approximately 22 + 2 oC. Ozone exposures will be conducted in a (6 ft x 6 ft x 8 ft) stainless steel chamber with a continuous supply of exposure medium. Ozone will be monitored continuously.
  Interventions: Other: Ozone exposure
- Diesel exhaust exposure (Other): Exposure to diesel exhaust will be conducted in an exposure chamber at the EPA Human Studies Facility on the UNC campus. Each subject will be exposed to diesel exhaust (up to 300 ug/m3). Subjects will begin exercising on an exercise bike. Each exercise session will consist of a 15 minute exercise interval at a level of up to 25 L/m2/BSA followed by a 15 minute rest period. The exposure atmosphere will be at approximately 40 + 10% RH and approximately 22 + 2 oC. The DE will be generated from a diesel generator used to power a load bank that is located outside the Human Studies Facility, and subsequently introduced into the exposure chamber after different dilutions with clean HEPA and charcoal filtered and humidified air to give a chamber concentration of up to 300 μg/m3.
  Interventions: Other: Diesel exhaust
- 18Ozone (Other): Exposure to ozone generated using the heavy non-radioactive isotope of oxygen (18O). Exposure to 0.3ppm 18O will be conducted in an exposure chamber at the EPA Human Studies Facility on the UNC campus. Each subject will be exposed for 2 hours. Subjects will begin exercising on an exercise bike. Each exercise session will consist of a 15 minute exercise interval at a level of up to 25 L/m2/BSA followed by a 15 minute rest period. The exposure atmosphere will be at approximately 40 + 10% RH and approximately 22 + 2 oC. Ozone exposures will be conducted in a (6 ft x 6 ft x 8 ft) stainless steel chamber with a continuous supply of exposure medium. Ozone will be monitored continuously.
  Interventions: Other: Ozone18

INTERVENTIONS:
Other: Ozone exposure — Exposure to 0.3ppm ozone for 2 hours
  Other Names: O3
  Arms: Ozone exposure
Other: Diesel exhaust — Diesel exhaust generated from a diesel generator delivered to the exposure at a target concentration of 300 μg/m3
  Other Names: DE; DEP
  Arms: Diesel exhaust exposure
Other: Ozone18 — Exposure to ozone generated using the heavy non-radioactive isotope of oxygen (18O).
  Other Names: O18
  Arms: 18Ozone
Other: Clean Air — Exposure to air which has been scrubbed to remove air pollutants including ozone and particles.
  Other Names: CA
  Arms: Clean air exposure

SUMMARY:
Purpose: The purpose of this protocol is to compare the genetic and epigenetic effects between diesel exhaust and ozone exposure in healthy individuals and in mild/moderate asthmatics.

Participants: The investigators will recruit up to 30 mild to moderate asthmatics and up to 50 healthy adults to participate in this study.

Procedures (methods): Subjects will be exposed to clean air, to 300 µg/m3 of diesel exhaust for 2 hours and to 0.3 ppm of ozone for 2 hours with intermittent exercise in a controlled environment chamber. Primary endpoints will include spirometry and lung cell changes post-exposure. Secondary endpoints will include analysis of blood clotting/coagulation factors, Holter monitoring of cardiac parameters, analysis of soluble factors present in plasma and bronchial lavage and analysis of intracellular factors present in lung tissue obtained from a brush biopsy.

DETAILED DESCRIPTION:
This study will compare the epigenetic responses of healthy adults and adults with mild asthma to diesel exhaust and ozone exposures. Up to fifty subjects will be recruited into the healthy adult group and up to thirty subjects into the mild to moderate asthmatic group. Both the normal healthy group and the asthmatic group will be randomly exposed to clean air, diesel exhaust and ozone with exposures separated by a minimum of two weeks followed by a bronchoscopy procedure 18-24 h post-exposure. Additionally, the healthy group will participate in a second arm of the study in which they will be randomly exposed to clean air and ozone only separated by a minimum of 2 weeks followed by a bronchoscopy procedure 1 h post-exposure. Responses of primary interest will include: 1) genetic and epigenetic changes 2) FEV1 as measured by spirometry, and 3) lung inflammation and cell changes as evaluated by bronchoalveolar lavage. The performance of these tests and procedures are considered essential to conducting the study. Exploratory endpoints will include: blood CBC and differential, fibrinogen and platelets, changes in IL 6 and IL 8 comparing pre-exposure with post-exposure values. Safety endpoints will include comparison of temperature, telemetry, respiratory rate, O2 saturation and symptoms scores for pre- and post-exposure, and at 18-24 hours post-exposure. All medical procedures will be performed by study personnel.

Up to an additional 15 healthy subjects will be recruited specifically to be exposed to ozone generated using the heavy non-radioactive isotope of oxygen (18O). There is no risk to the subject of inhaling this isotope, which is naturally occurring in small concentrations. We have previously used 18Ozone in a study approved by the UNC IRB in 1993. The purpose of these exposures is to measure the amount of 18O label attached to airway epithelial cells removed during bronchoscopy and thus calculate the dose of ozone these cells received. We will draw a small blood sample but no other tests will be performed on these subjects other than routine spirometry to ensure they are not at risk for bronchoscopy.

Physical Examination Day:

Prior to recruitment into the study, subjects will undergo a physical exam. During this visit, a short review of the subject's history will be performed and vital signs, height and weight will be assessed (temperature, pulse, respiratory rate, and blood pressure), to determine whether the individual meets any major exclusion criteria for the study. Up to 50 ml of blood may be collected for a CBC/ differential, chemistry and lipid panels. At this time the subject may undergo a physical examination for bronchoscopy or may be scheduled for one at another time.

In order to participate in this study, subjects will be asked to:

* Avoid smoke and fumes for 24 hours before all visits.
* Avoid drinking alcohol 24 hours before all visits.
* Avoid strenuous exercise for 24 hours prior to and after all visits.
* No caffeine for 12 hours prior to all study visits.
* Eat a normal breakfast prior to the exposures where the bronchoscopy is being performed ~24 h post-exposure.
* Not eat or drink anything after midnight the night before the bronchoscopy. This includes not eating or drinking prior to the exposures in which the bronchoscopy is being performed 1 h post-exposure.

Training Day

1. Eligible subjects will report to the research lab for an approximate 2-hour training session.
2. Informed consent will be obtained.
3. Assessment of vital signs (temperature, pulse, respiratory rate, and blood pressure), oxygen saturation
4. Pregnancy tests will be administered to any women who may have child-bearing potential.
5. Subjects will be trained on the cycle ergometer and the work load to elicit a minute ventilation normalized for body surface of 25L/m2/BSA will be determined. In most subjects this will be about 50 L/minute (IE. VO2 of approximately 2.0 L/m). A cycle ergometer work setting of 75 to 100 watts will usually achieve such a physiological response
6. Subjects will perform spirometry.
7. Subjects will be shown chamber where exposures will take place. Study Arm 1 - Bronchoscopy ~24 h Post-Exposure (Healthy & Asthmatic Subjects)

Exposure Day 1

The subjects will be exposed to ozone, diesel exhaust and clean air on three separate occasions, with the exposures separated by a minimum of two weeks (these will be 2-visit exposure sessions). Subjects receiving 18Ozone, will only be exposed to ozone.

1. Subjects will be asked to arrive at the study site no sooner than 8 AM and will undergo assessment of vital signs (temperature, pulse, respiratory rate, and blood pressure), oxygen saturation, and symptom score assessment.
2. Pregnancy tests will be administered to any women who may have child-bearing potential.
3. A telemetry unit will be attached for cardiac monitoring.
4. Subject will be fitted with a Holter monitor and the subject will be asked to recline in a quiet dark place for 30 minutes. After approximately 20 minutes a time marker will be activated so that heart rate variability frequency readings can be taken over the next 10 minutes. The subject will wear the Holter monitor for the next 24 hrs. Subjects exposed to 18Ozone will not be fitted with a Holter.
5. Venipuncture: Up to 80 ml of blood will be collected for a CBC/ differential, and may be used for assessment of coagulation function and markers, phagocytic function, inflammation, and cell surface markers. A portion of the sample may be used for RNA isolation for microarray analysis and for DNA isolation for genotyping purposes. Pre-exposure blood will not be taken from subjects being exposed to 18Ozone
6. Baseline Spirometry
7. Exposure sessions: Exposure to ozone, diesel exhaust or clean air will be conducted in an exposure chamber at the EPA Human Studies Facility on the UNC campus. Each subject will be exposed up to 0.3ppm ozone, diesel exhaust (up to 300 ug/m3) or clean air for 2 hours. Subjects will begin exercising on an exercise bike. Each exercise session will consist of a 15 minute exercise interval at a level of up to 25 L/m2/BSA followed by a 15 minute rest period. Minute ventilation may be measured during each exercise period. Continuous heart rate and rhythm, and oxygen saturation, will be monitored using telemetry and pulse oximetry respectively. Blood pressure may be monitored intermittently. Subjects will be asked to refrain but not prohibited from using inhaled bronchodilator during exposures; if medication use is necessary subjects will be instructed to maintain consistent medication use across the two exposures. The subjects will be able to end their exposure and exit the chamber at any time. Indications for terminating the exposure include significant respiratory distress or dyspnea, chest or angina-like pain, significant cardiac arrhythmias, pallor, ataxia, or a greater than 5 point drop in saturated oxygen (or a drop to lower than 89%). They will be monitored continuously by trained personnel and a physician is on call whenever a subject is undergoing a procedure at the facility. A detailed description of the physical facilities in the Human Studies Division of the U.S. EPA Health Effects Research Laboratory located on the UNC-CH campus have been published as U.S. Government Publication EPA-600/1-78-064, and is on file in the office of the UNC Committee on the Protection of the Rights of Human Subjects. The medical station of the Human Studies Division includes a fully-equipped medical examination room, a cardiac/respiratory emergency cart, a subject recovery room, a nurse's station, a waiting room and conference rooms. The facility is staffed by qualified RNs, and an on-site physician is available to respond to a medical emergency in a timely manner. The exposure atmosphere will be at approximately 40 + 10% RH and approximately 22 + 2 oC. The DE will be generated from a diesel generator used to power a load bank that is located outside the Human Studies Facility, and subsequently introduced into the exposure chamber after different dilutions with clean HEPA and charcoal filtered and humidified air to give a chamber concentration of up to 300 μg/m3. The monitoring analyzer registers a concentration in real time. Exposures will be terminated at values ≥ 400 µg/m3 during runs in which the exposure targets 300 µg/m3 DE. This safety limit will prevent an inhalational exposure greater than 1080 µg, which assumes that the subject will inhale 2.7 m3 during the 120 min exposure. Levels of carbon monoxide (CO), and oxides of nitrogen (NOx; mainly NO, and some NO2), will be kept under 10 ppm CO, 15 ppm NO, and 2.5 ppm NO2 or the exposure will be terminated. [The OSHA 8 hr time-weighted average (TWA) for these substances are: CO=50 ppm; NO=25 ppm; NO2=5 ppm; Diesel fuel used for the study will be purchased as a commercial ultra low sulfur fuel. Subjects will enter the exposure chamber (about 6 ft x 6 ft x 8 ft ). Particle mass will be measured in real time. Particle size distribution may not be determined during each subject exposure but at regular intervals (e.g., monthly) to show that the size distribution does not change radically. Filter samples will also be analyzed for chemical composition of particles. Ozone exposures will be conducted in a (6 ft x 6 ft x 8 ft) stainless steel chamber with a continuous supply of exposure medium. Ozone will be monitored continuously. Immediately post exposure, subjects will again undergo spirometry, Holter monitor frequency reading, symptom scoring and assessment of vital signs.
8. Then, up to 80 ml of blood will be collected for a CBC/ differential, assessment of coagulation function, blood leukocyte phagocytic function, cytokines, cell surface markers and RNA isolation for microarray analysis. Subjects exposed to 18Ozone will have only 20 mls of blood removed for analysis of 18O tag present on blood cells and have post exposure Spirometry measurements.
9. Subjects exposed to 18Ozone will have bronchoscopy performed about 1 hr post-exposure.

   Exposure to 18Ozone and undergoing a bronchoscopy approximately one hour later should not increase the risk to the subjects. We have completed two earlier studies in which subjects underwent bronchoscopy following exposure to concentrations of ozone higher than used in this study, and encountered no problems. Others have also published studies in which subjects were exposed to ozone followed by bronchoscopy one hour later
10. Subjects will then be assessed and discharged by the nursing staff.

Exposure Day 2 (approximately 24 hours after exposure) Subjects being exposed to 18O will not be returning for a Day 2

The subject will arrive at the U.S. EPA HSF for:

1. Vital sign monitoring.
2. Symptom scoring.
3. Venipuncture: up to 80 ml of blood will be collected for a CBC/ differential, coagulation function, assessment of blood monocyte phagocytic function, inflammation, and cell surface markers, and RNA isolation for microarray analysis.
4. Holter monitor frequency reading and removal
5. Spirometry
6. Bronchoscopy. Subjects will have undergone a physical examination including assessment for suitability for transnasal fiberoptic bronchoscopy at the Human Studies Facility by a board certified or board eligible pulmonologist.

Prior to the procedure, subjects will perform spirometry (as above); bronchoscopy will not be performed if lung function does not meet the recommended performance level (NIH guidelines; FEV1≥ 60 % predicted). Prior to bronchoscopy, a small tube (IV) will be placed in a vein for potential use in administering fluids. Subjects will receive inhaled albuterol prior to the bronchoscopy at the discretion of the pulmonary physician performing the procedure. Bronchoscopy with bronchoalveolar lavage and brush biopsy will be performed by a licensed physician who is Board certified or board eligible in pulmonary medicine and is experienced in fiberoptic bronchoscopy. The physician will be assisted by at least one R.N experienced in bronchoscopy. The subjects will be monitored closely throughout the procedure in the following manner: 1) Chest electrodes for continuous electrocardiogram, 2) Pulse oximetry of arterial blood, and 3) blood pressure monitoring using an electronic sphygmomanometer. Subjects may be premedicated with IV atropine (0.6 mg) to prevent bradycardia and hypotension that could result from vagal stimulation provoked by passing the bronchoscope through the subject's larynx and to minimize the amount of airways secretions. Nasal oxygen will be administered during the procedure. No sedatives and/or narcotics are administered at any time during bronchoscopy. We have found that premedication with sedatives (midazolam) or with opiates (demerol) is not required for research bronchoscopy subjects. Avoidance of these drugs reduces procedure risk and markedly shortens post-procedure recovery time. Neosynephrine will be used to decongest nasal passages, followed by gargling with a lidocaine solution for a few seconds to anesthetize the throat. The subject will then sniff (snort) a small amount of lidocaine jelly through one nostril to anesthetize the nose and the back of throat. A Q-tip with lidocaine jelly will be gently inserted into the nose to ensure that it is completely numb before the bronchoscope is inserted. Topical lidocaine anesthesia will be administered to the larynx and lower airways through the bronchoscope for subject comfort and to prevent cough, with a maximum dose of 15 ml of 2% lidocaine solution (360 mg lidocaine) Up to 8 endobronchial brush biopsies will be obtained from the lower trachea and right and left mainstem bronchi. A cytology brush (Bronchoscope Cytology Brush; Bard, Tewksbury, MA) is applied to the region under direct visualization. For a single brushing, six passes, each with a linear excursion of approximately 2-5 cm, are made with the brush along the endobronchial surface. Bronchoalveolar lavage will be performed in the right middle lobe using a total volume of up to 250 cc of sterile 0.9% saline; from one to 5 aliquots of 50 cc each will be injected and immediately aspirated through the channel in the bronchoscope using a syringe.

Subjects are observed and monitored for a minimum of 1 to 2 hours after the procedure in the on-site medical station by a registered nurse with physician supervision. At discharge subjects will be symptom-free. At least 2 physicians, including the responsible bronchoscopist, will be available (24 hours daily) to subjects who develop any symptoms after discharge. The subject is discharged by a physician and is provided with the names and telephone numbers of the bronchoscopist and one other physician. The subject is contacted 24 hours post-bronchoscopy to ask about any untoward effects.

Subjects will return to the U.S. EPA HSF for an additional exposure sessions and post exposure bronchoscopies (air control, ozone or diesel exhaust) after a minimum time interval of two weeks.

Study Arm 2 - Bronchoscopy 1 h Post-Exposure (Healthy Subjects ONLY)

Exposure Day 1

The subjects will be exposed to ozone and clean air on two separate occasions, with the exposures separated by a minimum of two weeks (these will be 1-visit exposure sessions).

1. Subjects will be asked to arrive at the study site no sooner than 8 AM and will undergo assessment of vital signs (temperature, pulse, respiratory rate, and blood pressure), and oxygen saturation.
2. Pregnancy tests will be administered to any women who may have child-bearing potential.
3. A telemetry unit will be attached for cardiac monitoring.
4. Baseline Spirometry
5. A saline lock will be placed in the subject's arm in preparation for IV fluids to be administered post-exposure.
6. Exposure sessions: Exposure to ozone or clean air will be conducted in an exposure chamber at the EPA Human Studies Facility on the UNC campus. Each subject will be exposed up to 0.3ppm ozone or clean air for 2 hours. Subjects will begin exercising on an exercise bike. Each exercise session will consist of a 15 minute exercise interval at a level of up to 25 L/m2/BSA followed by a 15 minute rest period. Minute ventilation may be measured during each exercise period. Continuous heart rate and rhythm, and oxygen saturation, will be monitored using telemetry and pulse oximetry respectively. Blood pressure may be monitored intermittently. The subjects will be able to end their exposure and exit the chamber at any time. Indications for terminating the exposure include significant respiratory distress or dyspnea, chest or angina-like pain, significant cardiac arrhythmias, pallor, ataxia, or a greater than 5 point drop in saturated oxygen (or a drop to lower than 89%). They will be monitored continuously by trained personnel and a physician is on call whenever a subject is undergoing a procedure at the facility. A detailed description of the physical facilities in the Human Studies Division of the U.S. EPA Health Effects Research Laboratory located on the UNC-CH campus have been published as U.S. Government Publication EPA-600/1-78-064, and is on file in the office of the UNC Committee on the Protection of the Rights of Human Subjects. The medical station of the Human Studies Division includes a fully-equipped medical examination room, a cardiac/respiratory emergency cart, a subject recovery room, a nurse's station, a waiting room and conference rooms. The facility is staffed by qualified RNs, and an on-site physician is available to respond to a medical emergency in a timely manner. The exposure atmosphere will be at approximately 40 + 10% RH and approximately 22 + 2 oC. Ozone exposures will be conducted in a (6 ft x 6 ft x 8 ft) stainless steel chamber with a continuous supply of exposure medium. Ozone will be monitored continuously. Immediately post exposure, subjects will again undergo spirometry and assessment of vital signs.
7. IV fluids will be administered prior to the bronchoscopy to ensure proper hydration of the subject
8. Subjects will have bronchoscopy performed about 1 hr post-exposure. Undergoing a bronchoscopy approximately one hour post-exposure should not increase the risk to the subjects. We have completed two earlier studies in which subjects underwent bronchoscopy following exposure to concentrations of ozone higher than used in this study, and encountered no problems. Others have also published studies in which subjects were exposed to ozone followed by bronchoscopy one hour later.

Subjects will have undergone a physical examination including assessment for suitability for transnasal fiberoptic bronchoscopy at the Human Studies Facility by a board certified or board eligible pulmonologist. Prior to the procedure, subjects will perform spirometry (as above); bronchoscopy will not be performed if lung function does not meet the recommended performance level (NIH guidelines; FEV1≥ 60 % predicted). Bronchoscopy with bronchoalveolar lavage and brush biopsy will be performed by a licensed physician who is Board certified or board eligible in pulmonary medicine and is experienced in fiberoptic bronchoscopy. The physician will be assisted by at least one R.N experienced in bronchoscopy. The subjects will be monitored closely throughout the procedure in the following manner: 1) Chest electrodes for continuous electrocardiogram, 2) Pulse oximetry of arterial blood, and 3) blood pressure monitoring using an electronic sphygmomanometer. Subjects may be premedicated with IV atropine (0.6 mg) to prevent bradycardia and hypotension that could result from vagal stimulation provoked by passing the bronchoscope through the subject's larynx and to minimize the amount of airways secretions. Nasal oxygen will be administered during the procedure. No sedatives and/or narcotics are administered at any time during bronchoscopy. We have found that premedication with sedatives (midazolam) or with opiates (demerol) is not required for research bronchoscopy subjects. Avoidance of these drugs reduces procedure risk and markedly shortens post-procedure recovery time. Neosynephrine will be used to decongest nasal passages, followed by gargling with a lidocaine solution for a few seconds to anesthetize the throat. The subject will then sniff (snort) a small amount of lidocaine jelly through one nostril to anesthetize the nose and the back of throat. A Q-tip with lidocaine jelly will be gently inserted into the nose to ensure that it is completely numb before the bronchoscope is inserted. Topical lidocaine anesthesia will be administered to the larynx and lower airways through the bronchoscope for subject comfort and to prevent cough, with a maximum dose of 15 ml of 2% lidocaine solution (360 mg lidocaine) Up to 8 endobronchial brush biopsies will be obtained from the lower trachea and right and left mainstem bronchi. A cytology brush (Bronchoscope Cytology Brush; Bard, Tewksbury, MA) is applied to the region under direct visualization. For a single brushing, six passes, each with a linear excursion of approximately 2-5 cm, are made with the brush along the endobronchial surface. Bronchoalveolar lavage will be performed in the right middle lobe using a total volume of up to 250 cc of sterile 0.9% saline; from one to 5 aliquots of 50 cc each will be injected and immediately aspirated through the channel in the bronchoscope using a syringe.

Subjects are observed and monitored for a minimum of 1 to 2 hours after the procedure in the on-site medical station by a registered nurse with physician supervision. At discharge subjects will be symptom-free and able to void urine. At least 2 physicians, including the responsible bronchoscopist, will be available (24 hours daily) to subjects who develop any symptoms after discharge. The subject is discharged by a physician and is provided with the names and telephone numbers of the bronchoscopist and one other physician. The subject is contacted 24 hours post-bronchoscopy to ask about any untoward effects.

Subjects will return to the U.S. EPA HSF for an additional exposure sessions and post exposure bronchoscopies (air control or ozone) after a minimum time interval of two weeks.

We anticipate performing several clinical procedures during the course of this study which include primary, secondary and exploratory endpoints. However, it is possible that not all procedures will be performed on every subject. If we are unable to perform a procedure, because of a investigator problem (such as but not limited too building/equipment failures, weather delays, or staffing issues), then the patient will be compensated for said procedure(s) and time on that day and may be rescheduled.

ELIGIBILITY:
Inclusion Criteria:

Healthy Individuals Specific Inclusion Criteria

1. Physical exams will be performed by study physicians during the screening visit (IRB approved EPA protocol 95-EPA-66).
2. Normal lung function (pre or post albuterol), defined by Knudson 1976/1984 as:

   - FVC of > 75 % of that predicted for gender, ethnicity, age and height.

   - FEV1 of > 75 % of that predicted for gender, ethnicity, age and height.

   - FEV1/FVC ratio of > 75 % of predicted values.
3. Oxygen saturation of > 96 %.
4. Ability to tolerate intervals of moderate exercise

Mild to Moderate Asthmatics

Inclusion Criteria:

1. Physical exams will be performed by study physicians during the screening visit (IRB approved EPA protocol 95-EPA-66) where diagnosis will be judged by EPA physicians.
2. Mild/Moderate asthmatics as defined by NHLBI guidelines.
3. Positive history of asthma (wheezing, chest tightness, and reversible airway obstruction);
4. Baseline FEV1/FVC ≥ 60%;
5. Oxygen saturation of ≥ 94%
6. Ability to tolerate moderate exercise

Exclusion Criteria:

* Healthy Individuals

  1. A history of chronic illnesses such as diabetes, rheumatological diseases, immunodeficiency state, known clinically significant cardiac disease (including myocardial infarction, congestive heart failure and angina), chronic respiratory diseases such as chronic obstructive pulmonary disease, and lung cancer.
  2. If the subject is pregnant, attempting to become pregnant or breastfeeding.
  3. Allergy to any medications which may be used or prescribed in the course of this study.
  4. Subjects currently taking mega doses of vitamins and supplements, homeopathic/naturopathic medicines or medications which may impact the results of the PM and/or ozone challenge or interfere with any other medications potentially used in the study (to include systemic steroids and beta blockers). Subjects must refrain from all over the counter anti-inflammatory agents including those for allergies, and naproxen, and anti-oxidants for a period of one week prior to exposure. Medications not specifically mentioned here may be reviewed by the investigators prior to a subject's inclusion in the study.
  5. Smoking history within 2 years of the study.
  6. Use of inhaled steroids, cromolyn, or leukotriene inhibitors (Montelukast, Zafirkulast, etc) initiated within the past month (except for use of cromolyn exclusively prior to exercise). Patients must be on a stable regimen of therapy.
  7. Untreated hypertension (> 150 systolic, > 90 diastolic)
  8. Dementia.
  9. Unspecified illnesses, which in the judgment of the investigator might increase the risk associated with PM inhalation challenge or exercise, will be a basis for exclusion.
  10. History of skin allergy to tape or electrodes.
  11. Subjects who do not understand or speak English
  12. Subjects who are unable to perform moderate exercise

      Exclusion criteria for bronchoscopy:

  <!-- -->

  1. Any food or fluids after midnight prior to bronchoscopy
  2. FEV1/FVC ratio less than 60% predicted on AM of bronchoscopy.
  3. Regular use of aspirin or other nonsteroidal anti-inflammatory drugs (which inhibit platelet function).

     Mild to Moderate Asthmatics

     Use of oral steroid therapy within the past month

  2. Physician directed emergency treatment for asthma exacerbation within the preceding 6 months.

  3. Abnormal EKG that precludes evaluating heart rate variability. 4. Aside from mild/moderate asthma, a history of chronic illnesses such as diabetes, rheumatological diseases, immunodeficiency state, known clinically significant cardiac disease (including myocardial infarction, congestive heart failure and angina), chronic respiratory diseases such as chronic obstructive pulmonary disease or severe asthma, and cancer (possible exception for history of nonmelanoma skin cancer).

  5. If the subject is pregnant, attempting to become pregnant or breastfeeding. 6. Allergy to any medications which may be used or prescribed in the course of this study 7. Subjects currently taking mega doses of vitamins and supplements, homeopathic/naturopathic medicines or medications which may impact the results of the PM challenge or interfere with any other medications potentially used in the study (to include systemic steroids and beta blockers). Subjects must refrain from all over the counter anti-inflammatory agents including those for allergies, and naproxen, and anti-oxidants for a period of one week prior to exposure. Medications not specifically mentioned here may be reviewed by the investigators prior to a subject's inclusion in the study.

  8. Dosing level of an inhaled steroid must be consistent with mild asthma as outlined by the NHLBI NAEPP guidelines. Regular use of oral corticosteroids, or use of inhaled steroid at doses typically used for severe asthma, will result in exclusion of that individual from the protocol.

  9. Severe asthmatics as defined by: nighttime symptoms of cough or wheeze greater than 1 time per week at baseline, daily exacerbation of asthma or requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness, but not to include prophylactic use of albuterol prior to exercise), more than mild interference with normal activity, any episode of physician directed emergency treatment for asthma requiring oral corticosteroid therapy within the past twelve months.

  10. Smoking history within 2 years of study. 11. Use of inhaled steroids, cromolyn, or leukotriene inhibitors (Montelukast, Zafirkulast, etc) initiated within the past month (except for use of cromolyn exclusively prior to exercise). Patients must be on a stable regimen of therapy.

  12. History of skin allergy to tape or electrodes. 13. History of respiratory diseases other than allergic rhinitis and asthma 14. Untreated hypertension (> 150 systolic, > 90 diastolic) 15. Dementia. 16. Unspecified illnesses, which in the judgment of the investigator might increase the risk associated with PM inhalation challenge or exercise, will be a basis for exclusion.

  17. Subjects who do not understand or speak English 18. Subjects who are unable to perform moderate exercise

Exclusion criteria for bronchoscopy:

1. Any food or fluids after midnight prior to bronchoscopy
2. FEV1/FVC ratio less than 60% predicted on AM of bronchoscopy.
3. Regular use of aspirin or other nonsteroidal anti-inflammatory drugs (which inhibit platelet function).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Airway responses | Pre exposure to 24hours post exposure
  Airway responses include spirometry and lung cell changes following exposure to either clean air, ozone or diesel exhaust Lung cell changes include change in number and type of cells, changes in genetic (gene expression) and epigenetic responses (primarily changes in DNA methylation, microRNA expression and chromatin modification.

SECONDARY OUTCOMES:
Cardiovascular responses | Pre exposure to 24hours post exposure
  Cardiovascular responses are analysis of blood clotting/coagulation factors and Holter monitoring of cardiac parameters following exposure to clean air, ozone or diesel exhaust
Soluble factors | Pre exposure to 24hours post exposure
  Analysis of soluble factors present in plasma and bronchial lavage and analysis of intracellular factors present in lung tissue obtained from a brush biopsy following exposure to clean air ozone or diesel exhaust

CONTACTS AND LOCATIONS:
Overall Officials: David Diaz-Sanchez, Ph.D., Study Director — U.S. Environmental Protection Agency; Kelly Duncan, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- U.S. EPA Human Studies Facility, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Sommer AJ, Okonkwo J, Monteiro J, Bind MC. A permutation-based approach using a rank-based statistic to identify sex differences in epigenetics. Sci Rep. 2023 Sep 8;13(1):14838. doi: 10.1038/s41598-023-41360-6. PMID 37684282
- [Derived] Miller DB, Ghio AJ, Karoly ED, Bell LN, Snow SJ, Madden MC, Soukup J, Cascio WE, Gilmour MI, Kodavanti UP. Ozone Exposure Increases Circulating Stress Hormones and Lipid Metabolites in Humans. Am J Respir Crit Care Med. 2016 Jun 15;193(12):1382-91. doi: 10.1164/rccm.201508-1599OC. PMID 26745856
- [Derived] Devlin RB, Duncan KE, Jardim M, Schmitt MT, Rappold AG, Diaz-Sanchez D. Controlled exposure of healthy young volunteers to ozone causes cardiovascular effects. Circulation. 2012 Jul 3;126(1):104-11. doi: 10.1161/CIRCULATIONAHA.112.094359. Epub 2012 Jun 25. PMID 22732313